CLINICAL TRIAL: NCT05709886
Title: A Prospective, Single-arm, Multicenter Clinical Trial of Safety and Effectiveness of Endoscopic Ultrasound-guided Laser Ablation for Liver Cancer by LaserPro Diode Laser System
Brief Title: A Prospective, Single-arm, Multicenter Clinical Trial of Safety and Effectiveness of EUS-LA for Liver Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Yiwu Central Hospital (Other); Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eusLAliver
Record Dates: First submitted 2023-01-25; First posted 2023-02-02 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-12

CONDITIONS: Liver Cancer
Keywords: liver cancer; laser; ablation; endoscopic ultrasound
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: To evaluate whether the LaserPro Diode Laser System under the guidance of EUS can achieve the safety and effectiveness of local ablation for liver cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS-LA by LaserPro Diode Laser System (Experimental): This trial is a prospective, single-arm, multi-center clinical trial. Four hospitals with national medical trial institution qualifications are selected as clinical trial centers. Qualified participants will receive endoscopic ultrasound (EUS)-guided laser ablation (LA) by LaserPro Diode Laser System according to the routine procedures. The results will be recorded according to the requirements of the primary and secondary efficacy indicators. After then, statistical comparisons of effectiveness and safety of the procedure will be made according to groups.
  Interventions: Device: EUS-LA by LaserPro Diode Laser System

INTERVENTIONS:
Device: EUS-LA by LaserPro Diode Laser System — This trial is a prospective, single-arm, multi-center clinical trial. Four hospitals with national medical trial institution qualifications are selected as clinical trial centers. Qualified participants will receive endoscopic ultrasound (EUS)-guided laser ablation (LA) by LaserPro Diode Laser System according to the routine procedures. The results will be recorded according to the requirements of the primary and secondary efficacy indicators. After then, statistical comparisons of effectiveness and safety of the procedure will be made according to groups.

SUMMARY:
This trial is a prospective, single-arm, multi-center clinical trial. Four hospitals with national medical trial institution qualifications are selected as clinical trial centers. Qualified participants will receive endoscopic ultrasound-guided laser ablation by LaserPro Diode Laser System according to the routine procedures. The results will be recorded according to the requirements of the primary and secondary efficacy indicators. After then, statistical comparisons of effectiveness and safety of the procedure will be made according to groups.

DETAILED DESCRIPTION:
The prospective, single-arm, multi-center clinical trial is to evaluate whether the endoscopic ultrasound (EUS)-guided laser ablation (LA) by LaserPro Diode Laser System can achieve the safety and effectivenessof liver cancer ablation treatment. Four hospitals with national medical clinical trial institution qualifications are selected as clinical trial centers. This clinical trial requires 69 subjects. Qualified participants will receive EUS-guided LA by LaserPro Diode Laser System according to the routine procedures. The results will be recorded according to the requirements of the primary outcome (the complete ablation (CA) rate and the effective rate of EUS-guided LA by LaserPro Diode Laser System for liver cancer) and secondary outcomes (technical success rate, major complication rate, partial response rate, secondary ablation rate, progression-free survival (PFS), overall survival rate (OS), local tumor progression (LTP), distant tumor recurrence (DTR), quality of life score and alpha-fetoprotein levels). The one-month follow-up after the operation, three-phase MRI, liver function and tumor markers were reviewed monthly to observe the lesion necrosis and tumor marker changes. After that, tumor markers, three-phase MRI of liver were examined every 2 to 3 months. After then, statistical comparisons of safety and effectivenessof the producedure will be made according to groups.

ELIGIBILITY:
Inclusion Criteria:

1. Liver malignant tumors with clear histopathology and cytology, or liver malignant tumors that meet clinical diagnosis and staging criteria.
2. Liver tumors within the scope of EUS scanning.
3. Single tumor≤ 3cm in diameter and the number of visible tumor were no more than 3. According to CT and MRI, there are no macrovascular and bile duct invasions visible by the naked eye.
4. Liver function: Child-Pugh A or B.
5. Age: 18-75 years old, regardless of gender.
6. Patients signed informed consent to participate in the trial.

Exclusion Criteria:

1. Contraindication for EUS or the target tumor were beyond the scope of EUS scanning.
2. Liver function: Child-pugh C, those could not improve after liver protective treatment.
3. Uncorrectable coagulation dysfunction and severe haematological abnormalities, who tend to severe bleeding; platelet count less than 50×109/L, prothrombin time more than 30s or prothrombin activity less than 40%.
4. Severe failure of major organs such as kidney, heart, lung and brain.
5. Uncontrolled infection in any organ, especially inflammation of the biliary system.
6. Esophageal (bottom of stomach) varices rupture and bleeding within 1 month before treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Complete ablation rate | 1 month
  Defined as the absence of any contrast uptake within or at the periphery of the ablative zone. One month after either one session or multiple LA sessions, CTA was confirmed by contrast-enhanced MRI.
Effectiveness analysis | 6 months
  The effective rate of EUS-LA by LaserPro Diode Laser System for liver cancer was evaluated by mRECIST criteria.

SECONDARY OUTCOMES:
Technical success rate | 1 month
  Technical success rate of EUS-LA by LaserPro Diode Laser System for liver cancer.
Major complication rate | 6 months
  Major complication rate after EUS-LA by LaserPro Diode Laser System for liver cancer.
Partial response rate | 6 months
  Partial response rate after EUS-LA by LaserPro Diode Laser System for liver cancer.
Secondary ablation rate | 6 months
  Secondary ablation rate after EUS-LA by LaserPro Diode Laser System for liver cancer.
Progression-free survival (PFS) | 6 months
  Progression-free survival after EUS-LA by LaserPro Diode Laser System for liver cancer.
Overall survival rate (OS) | 6 months
  Overall survival rate after EUS-LA by LaserPro Diode Laser System for liver cancer.
Local tumor progression (LTP) | 6 months
  Local tumor progression after EUS-LA by LaserPro Diode Laser System for liver cancer.
Distant tumor recurrence (DTR) | 6 months
  Distant tumor recurrence after EUS-LA by LaserPro Diode Laser System for liver cancer.
Quality of life score | 6 months
  Quality of life score of participants after EUS-LA by LaserPro Diode Laser System for liver cancer.
Alpha-fetoprotein levels | 6 months
  The alpha-fetoprotein levels of participants after EUS-LA by LaserPro Diode Laser System for liver cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Tian'an Jiang, PhD, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Nault JC, Sutter O, Nahon P, Ganne-Carrie N, Seror O. Percutaneous treatment of hepatocellular carcinoma: State of the art and innovations. J Hepatol. 2018 Apr;68(4):783-797. doi: 10.1016/j.jhep.2017.10.004. Epub 2017 Oct 13. PMID 29031662
- [Background] Hong K, Georgiades CS, Geschwind JF. Technology insight: Image-guided therapies for hepatocellular carcinoma--intra-arterial and ablative techniques. Nat Clin Pract Oncol. 2006 Jun;3(6):315-24. doi: 10.1038/ncponc0512. PMID 16757969
- [Background] Villanueva A. Hepatocellular Carcinoma. N Engl J Med. 2019 Apr 11;380(15):1450-1462. doi: 10.1056/NEJMra1713263. No abstract available. PMID 30970190
- [Background] Petrowsky H, Fritsch R, Guckenberger M, De Oliveira ML, Dutkowski P, Clavien PA. Modern therapeutic approaches for the treatment of malignant liver tumours. Nat Rev Gastroenterol Hepatol. 2020 Dec;17(12):755-772. doi: 10.1038/s41575-020-0314-8. Epub 2020 Jul 17. PMID 32681074
- [Background] Pacella CM, Francica G, Di Lascio FM, Arienti V, Antico E, Caspani B, Magnolfi F, Megna AS, Pretolani S, Regine R, Sponza M, Stasi R. Long-term outcome of cirrhotic patients with early hepatocellular carcinoma treated with ultrasound-guided percutaneous laser ablation: a retrospective analysis. J Clin Oncol. 2009 Jun 1;27(16):2615-21. doi: 10.1200/JCO.2008.19.0082. Epub 2009 Mar 30. PMID 19332729
- [Background] Arienti V, Pretolani S, Pacella CM, Magnolfi F, Caspani B, Francica G, Megna AS, Regine R, Sponza M, Antico E, Di Lascio FM. Complications of laser ablation for hepatocellular carcinoma: a multicenter study. Radiology. 2008 Mar;246(3):947-55. doi: 10.1148/radiol.2463070390. Epub 2008 Jan 14. PMID 18195382
- [Background] Di Costanzo GG, Tortora R, D'Adamo G, De Luca M, Lampasi F, Addario L, Galeota Lanza A, Picciotto FP, Tartaglione MT, Cordone G, Imparato M, Mattera S, Pacella CM. Radiofrequency ablation versus laser ablation for the treatment of small hepatocellular carcinoma in cirrhosis: a randomized trial. J Gastroenterol Hepatol. 2015 Mar;30(3):559-65. doi: 10.1111/jgh.12791. PMID 25251043
- [Background] Di Costanzo GG, Francica G, Pacella CM. Laser ablation for small hepatocellular carcinoma: State of the art and future perspectives. World J Hepatol. 2014 Oct 27;6(10):704-15. doi: 10.4254/wjh.v6.i10.704. PMID 25349642
- [Background] Pacella CM, Francica G, Di Costanzo GG. Laser ablation for small hepatocellular carcinoma. Radiol Res Pract. 2011;2011:595627. doi: 10.1155/2011/595627. Epub 2011 Dec 4. PMID 22191028
- [Background] Chai W, Zhao Q, Song H, Cheng C, Tian G, Jiang T. Treatment response and preliminary efficacy of hepatic tumour laser ablation under the guidance of percutaneous and endoscopic ultrasonography. World J Surg Oncol. 2019 Aug 5;17(1):133. doi: 10.1186/s12957-019-1677-6. PMID 31383020
- [Background] Di Matteo F, Grasso R, Pacella CM, Martino M, Pandolfi M, Rea R, Luppi G, Silvestri S, Zardi E, Costamagna G. EUS-guided Nd:YAG laser ablation of a hepatocellular carcinoma in the caudate lobe. Gastrointest Endosc. 2011 Mar;73(3):632-6. doi: 10.1016/j.gie.2010.08.019. Epub 2010 Oct 27. No abstract available. PMID 21030019
- [Background] Jiang TA, Deng Z, Tian G, Zhao QY, Wang WL. Efficacy and safety of endoscopic ultrasonography-guided interventional treatment for refractory malignant left-sided liver tumors: a case series of 26 patients. Sci Rep. 2016 Dec 13;6:36098. doi: 10.1038/srep36098. PMID 27958384
- [Background] Jiang T, Tian G, Bao H, Chen F, Deng Z, Li J, Chai W. EUS dating with laser ablation against the caudate lobe or left liver tumors: a win-win proposition? Cancer Biol Ther. 2018 Mar 4;19(3):145-152. doi: 10.1080/15384047.2017.1414760. Epub 2018 Jan 25. PMID 29303406